CLINICAL TRIAL: NCT01804699
Title: Canadian National Arrhythmogenic Right Ventricular Cardiomyopathy
Brief Title: National ARVC Data Registry and Bio Bank
Acronym: ARVCRegistry
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Population Health Research Institute (Other); Medtronic (Industry); Boston Scientific Corporation (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Andrew Krahn, Professor, University of British Columbia
Other Study IDs: H12-03189
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: ARVC, Cardiomyopathy
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — If the participant consents to the biobanking arm of the study an additional blood sample (Please see the ARVC Lab Manual for details) will be collected at baseline and stored for subsequent analysis. These analyses may include measurement of serum Troponin T, NT-pro-BNP, C-reactive protein and other biomarkers to determine their association with the progression of disease; both in terms of cardiac structure (i.e. change in right ventricular volume) and electrical substrate (i.e. number of ICD shocks) over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proband: Probands - Participants diagnosed with ARVC according to the 2010 Task Force Criteria
- Family: First Degree Family member (blood related mother, father, sister, brother, child) of the proband

SUMMARY:
Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is an inherited condition that may cause life threatening irregular heart rhythms that often manifest as unexpected cardiac arrest or sudden death in early adulthood. The condition is difficult to diagnose and often is not noticed until a family member suffers a cardiac arrest or death.

The Canadian National ARVC registry will collect data from Inherited Heart Rhythm Clinics across Canada.

STUDY OBJECTIVES:

Primary:

1. To determine the natural history of ARVC (short/intermediate term), including risk of symptomatic arrhythmias and sudden death, for patients with the phenotype and those gene positive patients without phenotype evidence of disease.
2. To understand risk factors for sudden death/appropriate ICD use in ARVC, including test characteristics/performance and their relationship to outcomes (ECG, Holter, signal averaged ECG, loop recorders, imaging, voltage mapping, T wave alternans, cardiac biopsy and biomarkers).
3. To establish a phenotype genotype correlation, including comparison of patients with disease causing mutations, variants of unknown significance (VUS) and Task Force Criteria (TFC) positive, gene negative patients

DETAILED DESCRIPTION:
BACKGROUND:

Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is a familial condition characterized by onset of life threatening ventricular arrhythmias in early adulthood, presenting with ventricular tachycardia, cardiac arrest or sudden death1. The disease is diagnosed with a wide range of tests that focus on imaging the right ventricle and assessing for ambient arrhythmia or abnormal electrical substrate.

These factors are collated into a score that forms the ARVC Task Force Criteria, known to be specific but not sensitive 2, 3. These criteria have been revised in 2010, introducing a broader and more quantitative approach to diagnosis including genetic testing results, intended to enhance sensitivity without reducing specificity 4. An online tool for Task Force Criteria calculation has been developed by the Principal Investigator that enables calculation in real time, with export to PDF and excel format, free for public use (http://qstatistic.com/pdg/public.php?rep=arvc_cri).These criteria take into account electrocardiographic and imaging findings, along with tissue analysis and family history. They account for findings from genetic testing, confounded in part by the unknown significance of a positive genetic test in the absence of a phenotype in a disease with variable penetrance and expressivity 2, 4-12. The disease is predominantly caused by defects in cell-cell adhesion.

PROJECT APPROVAL PROCESS: For new projects and further analysis

New projects and proposals for the Canadian National ARVC Registry will be reviewed on a case-by-case basis by the Steering Committee. The following items must be included with each new proposal:

1. Project description with necessary background, hypotheses and methodology/protocol
2. A comprehensive list of funding source(s) with a detailed budget
3. Local Research Ethics Board (REB) approval

PATIENT RECRUITMENT & SCREENING PROCESS:

1. Patients will be approached to participate in the Registry in specialty clinics who are involved in the Registry across Canada.
2. Once informed consent is obtained ARVC affected patients will undergo baseline data collection including:

   1. Collection of standard clinical testing for ARVC (if affected patient) according to local clinical practice i.e. MRI, ECG etc. Family members will undergo screening as deemed necessary by the local investigator
   2. Baseline clinical history
   3. Family history and exercise history
   4. A family pedigree will be constructed.
   5. An online tool for pedigree construction has been developed by the Principal Investigator Dr. Andrew Krahn that enables creation of pedigrees in real time as well as the linking of patients in a genetics database, with export to PDF format, (demonstration version at https://ocrr.ca/pdg/i.php?loc=dmo, contact kgibbs@providencehealth.bc.ca for access)
   6. Patients will be enrolled in the database as prevalent cases that were previously identified, or incident cases
   7. Other testing if applicable
3. Genetic Information (if applicable). Once informed consent has been obtained patients will undergo baseline data collection and will be invited to participate in the optional DNA biobanking arm of the study
4. Genetic Screening for ARVC is a standard clinical evaluation for individuals with ARVC as well as their 1st degree family members this will be done clinically and sent to commercial laboratories as per the standard at each of the enrolling centres
5. If the participant consents to the biobanking arm of the study an additional blood sample (Please see the ARVC Lab Manual for details) will be collected at baseline and stored for subsequent analysis. These analyses may include measurement of serum Troponin T, NT-pro-BNP, C-reactive protein and other biomarkers to determine their association with the progression of disease; both in terms of cardiac structure (i.e. change in right ventricular volume) and electrical substrate (i.e. number of ICD shocks) over time.

DATA COLLECTION:

Baseline:

1. Patients will be required to provide written informed consent to participate in the study.
2. The local Research Ethics Board (REB) must approve all informed consent documents.
3. All demographic information, clinical testing and genetic results will be entered into a password-protected database.

Core Data Set (required):

The core data set consists of baseline and follow-up clinical testing that will establish participant eligibility according to 2010 Revised Task Force Criteria. The core data set will include the following:

1. Resting ECG
2. Signal averaged ECG
3. Transthoracic echocardiogram
4. Treadmill exercise test
5. 24 hour Holter monitor
6. Cardiac MRI

Additional test results (if clinically indicated):

The following comprises a typical list of additional test results that may be collected if available. These test results can be collected if they are clinically indicated for the participant(s).

1. Right ventricular angiography
2. Right ventricular biopsy
3. Right ventricular voltage map
4. Ability to induce ventricular tachycardia at Electrophysiologic testing
5. Transesophageal echocardiogram
6. T wave alternans
7. Cardiac CT scan

Genetic Testing and Results:

1. Optional blood drawn for banking at PHRI will be processed at each local site and shipped in Cryovials for banking at PHRI in Hamilton, Ontario. Specimen(s) collected (i.e. blood, saliva, DNA) will be processed locally before shipping to PHRI.
2. Blood drawn for standard clinical ARVC genetic testing at commercial laboratories in Canada (For example: in Ontario both SickKids Department of Paediatric Laboratory Medicine and CHEO Molecular Genetics Diagnostic Laboratory perform ARVC testing) can be packaged and shipped according to each of the local sites labs independent specifications.
3. Genetic testing results will be entered into a secure, password-protected database. These results are further de-identified with a code list so that there is no linkage to clinical data.

Follow-up:

Follow-up visits for the Registry will occur on an annual basis with the following testing:

1. Resting ECG
2. Signal averaged ECG
3. 24 hour Holter Monitor
4. Clinical History
5. Screening for any new cardiac symptoms, such as: syncope, palpitations, cardiac arrest, ICD implant, ICD therapy and sudden death

Clinical follow-up data will be collected according to standard local practice. It is ideal to reassess participants clinically, however if this is not feasible for some reason - a telephone interview can be conducted to assess any new clinical findings or new events that have taken place.

If the site wishes to conduct a telephone follow up - the following clinical testing is still required for the annual follow up visit:

1. Resting ECG
2. Signal averaged ECG if possible
3. 24 hour Holter Monitor

ECGs and Holter tracings can be obtained from remote areas and the findings entered into the database for annual follow up purposes.

3-Year Reassessment:

After 3 years participation in the study, participants will be reassessed based on the 2010 task force criteria. This includes the following:

1. Resting ECG
2. Signal averaged ECG
3. Transthoracic echocardiogram
4. Treadmill exercise test
5. 24 hour Holter monitor
6. Cardiac MRI
7. Clinical History
8. Screening for any new cardiac symptoms, such as: syncope, palpitations, cardiac arrest, ICD implant, ICD therapy and sudden death

There is currently no obligation to enter data beyond the 3 year mark, however sites are encouraged to continue follow up for participants indefinitely. The Registry is open-ended and with local REB approval participant's follow up data can continue to be entered as long as it is declared in the letter of information originally given to the participant.

DATA MANAGEMENT:

Data points for collection are present in the internet based database (see online demo at https://www.qstatistic.com/arvc/demo ). The database is hosted on the University of British Columbia Research Institute Vancouver British Columbia. The research institute is in compliance with national Canadian PIPEDA privacy guidelines. Data will be entered directly into the e-CRFs for electronic submission to a server located at UBC Research Institute,Vancouver BC and will not collect any personal identifiers (password protected internet based system).

Personal identifiers will not be collected and subject confidentiality will be further ensured in addition to maintaining de-identification by utilizing subject identification code numbers to correspond to data in the computerized files. Original files containing patient information will remain on file with the participating Investigator.

Individual subject medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited except for the following reason; medical information may be given to the subject's personal physician or to other appropriate medical personnel responsible for the subject's welfare. The eCRF (electronic clinical research form) system works best in the Internet browser Firefox©. This Internet browser can be downloaded from www.mozilla.org.

Access to the eCRFs will be issued once the site has local Ethics approval. .

ETHICAL CONSIDERATIONS

This trial will be conducted in compliance with the protocol, principles laid down in the Declaration of Helsinki, Good Clinical Practice (GCP), as defined by the International Conference on Harmonization (ICH), where applicable, and all other local regulatory requirements. Before study initiation, the enrolling site Investigator must have written and dated approval/favorable opinion from the Institutional Review Board/Independent Ethics Committee (IRB/IEC) for the protocol, and consent form.

ELIGIBILITY:
Inclusion Requirements:

1. 2010 Revised Task Force Criteria positive patients (please refer to Appendix 3.0)
2. 2010 Revised Task Force Criteria borderline patients
3. Disease causing ARVC pathogenic mutation* carriers with no TFC criteria for ARVC
4. Variants of unknown significance carriers with ≥1 minor TFC criterion
5. Age ≥ 2 years
6. First-degree relatives of 2010 Revised Task Force Criteria positive or borderline patients
7. Able and willing to provide informed consent, or has a parent/guardian able and willing to provide informed consent and/or able to sign an assent form

   * A pathogenic mutation is a DNA alteration associated with ARVC/D that alters or is expected to alter the encoded protein in a significant way, is unobserved or rare in a large non-ARVC/D control population, and either alters or is predicted to alter the structure or function of the protein (by computational (in silico) predictions and/or functional validation in a biological model system) or has demonstrated linkage to the disease phenotype in a conclusive pedigree 4. Mutation carriers by definition have a single major Task Force criterion.

EXCLUSION CRITERIA:

Exclusion Requirements:

1. Known condition that mimics ARVC - sarcoidosis (biopsy proven or with lung involvement), familial dilated cardiomyopathy not compatible with an ARVC variant, hypertrophic cardiomyopathy
2. Known inherited condition that predisposes to sudden death - Long or Short QT Syndrome, Catecholaminergic Polymorphic Ventricular Tachycardia and Brugada Syndrome
3. Age < 2 years
4. Life expectancy less than 1 year
5. Unable and/or unwilling to provide informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be identified from centers that form the Canadian Genetics Heart Rhythm (CGHR) Network of Inherited Heart Rhythm Clinics across Canada 25 (http://www.heartrhythmresearch.ca/).
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Natural History of ARVC | Three years
  To determine the natural history of ARVC (short/intermediate term), including risk of symptomatic arrhythmias and sudden death, for patients with the phenotype and those gene positive patients without phenotype evidence of disease.

SECONDARY OUTCOMES:
Risk Factors and Sudden Death | Three Years
  To understand risk factors for sudden death/appropriate ICD use in ARVC, including test characteristics/performance and their relationship to outcomes (ECG, Holter, signal averaged ECG, loop recorders, imaging, voltage mapping, T wave alternans, cardiac biopsy and biomarkers).

OTHER OUTCOMES:
Establishing a phenotype genotype correlation | Three Years
  To establish a phenotype genotype correlation, including comparison of patients with disease causing mutations, variants of unknown significance (VUS) and Task Force Criteria (TFC) positive, gene negative patients

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krahn, MD, Principal Investigator — University of British Columbia, Dept of Medicine, Head of Cardiology
Locations (16):
- Canada (16):
  - Libin Cardiovascular Institute of Alberta, University of Calgary, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - University of British Columbia, St. Paul's Hospital, Vancouver, British Columbia
  - University of Victoria, Victoria Jubilee Hospital, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II, Halifax Infirmary, Halifax, Nova Scotia
  - McMaster University, Faculty of Health Sciences, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - St. Justine Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie, Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No